CLINICAL TRIAL: NCT04704817
Title: Prospective Database for Colonic or Rectal Resection Surgery Patients
Acronym: CHIRCOLREC
Status: Not yet recruiting | Type: Observational
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: CHIRCOLREC-IPC 2018-017
Record Dates: First submitted 2021-01-08; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: obsevation — prospective data collection for colonic or rectal surgery

SUMMARY:
Colorectal cancer is the third most common cancer in men, after prostate and lung cancer. It represents 11.2% of all new cases of male cancer. In women, this cancer is the second most common after breast cancer (11.3% of all new cases of female cancer).

DETAILED DESCRIPTION:
Colorectal cancer is the second leading cause of cancer death in France. It accounts for nearly 12% of all cancer deaths, especially among those 65 and over. However, mortality has declined steadily since 1980.

Access to screening for colorectal cancer and resection of precancerous lesions partly explains this decline. All sexes combined, it is estimated that about one in five colorectal cancer is diagnosed at a limited local stage. The treatment is then less heavy and gives better results.

With the development of Enhanced Recovery After Surgery (ERAS) protocols and their extension to rectal excision, it becomes imperative to be able to collect operative data from these patients on a perennial basis for the purpose of evaluating our results. Finally, the evaluations resulting from this database could have prognostic value and ultimately allow us to adapt the surgical management of the patient according to the results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients treated for colonic and / or rectal resection in the oncological digestive surgery department of the Paoli-Calmettes Institute,
2. Patients over 18 years old,
3. Affiliation to a social security scheme, or beneficiary of such a scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adults treated ot to be treated for colonic and or rectal resection
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2051-03 (Estimated); Study Completion 2071-12 (Estimated)

PRIMARY OUTCOMES:
clinical events | 5 years
  to asses postoperative effects of colonic or rectal excision by collecting clinical events

IPD SHARING:
Plan to Share IPD: No